CLINICAL TRIAL: NCT05567614
Title: Platelets Indices and Its Role to Predict Liver Fibrosis in Patients With Chronic Hepatitis B Infection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Wafaa Adel Abdelghany, Platelets indices and its role to predict liver Fibrosis in patients with chronic hepatitis B infection, Assiut University
Other Study IDs: Platelets and liver fibrosis
Record Dates: First submitted 2022-10-02; First posted 2022-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Fibrosis, Liver
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 75: patients with chronic hepatitis B infection will be collected and underwill liver fibroscan then corelate between platelets indicies and predict degree of liver fibrosis
  Interventions: Radiation: Liver Fibroscan

INTERVENTIONS:
Radiation: Liver Fibroscan — Patients with CHB virus will do liver fibroscan and correlat between platelets count and degree of liver fibrosis
  Other Names: Elastography and Fibroscan

SUMMARY:
Platelets indices and its role to predict liver Fibrosis in patients with chronic hepatitis B infection

DETAILED DESCRIPTION:
Patients with chronic Hepatitis B infection will be collected and will do liver fibroscan to predict the degree of liver Fibrosis and correlate between the role of platelets count and degree of liver Fibrosis in patients with Chronic hepatitis B virus

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 70 years
* without a history of clinical illness

Exclusion Criteria:

* with other hepatitis virus infection; (b) with alcoholic liver disease; (c) with any disease related to fibrosis (such as connective tissue diseases, chronic obstructive pulmonary disease, kidney failure, tumors, and so on); (d) have received any anti-fibrosis therapy; and (e) pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients at Age from 18 to 70 years with chronic hepatits B infection will do liver fibroscan and correlate between platelets indicies and degree of liver fibrosis
  -
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2022-10-20 (Estimated); Primary Completion 2023-08-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Platelets indices and its role to predict liver Fibrosis in patients with chronic hepatitis B infection | Two years
  Correlation between platelets count and degree of liver Fibrosis in patients with chronic hepatitis B virus through liver fibroscan

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed AB Maghraby, Professor, Study Director — Assiut University
Locations (1):
- AssiutU, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No
the value of platelets count in evaluating the degree of liver fibrosis in patients with chronic hepatits B infecion

REFERENCES:
- [Background] Zhong LK, Zhang G, Luo SY, Yin W, Song HY. The value of platelet count in evaluating the degree of liver fibrosis in patients with chronic hepatitis B. J Clin Lab Anal. 2020 Jul;34(7):e23270. doi: 10.1002/jcla.23270. Epub 2020 May 4. PMID 32363594
- [Background] Tan YW, Zhou XB, Ye Y, He C, Ge GH. Diagnostic value of FIB-4, aspartate aminotransferase-to-platelet ratio index and liver stiffness measurement in hepatitis B virus-infected patients with persistently normal alanine aminotransferase. World J Gastroenterol. 2017 Aug 21;23(31):5746-5754. doi: 10.3748/wjg.v23.i31.5746. PMID 28883700